CLINICAL TRIAL: NCT02163746
Title: A Prospective, Randomized, Controlled Clinical Trial Comparing the Efficacy Carbon Dioxide (CO2) Laser Excision Versus Surgical Deroofing in the Treatment of Hidradenitis Suppurativa
Brief Title: Study to Compare Two Treatments for Axillary Hidradenitis Suppurativa: Carbon Dioxide Laser Versus Surgical Deroofing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Senior Staff Physician, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8606
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Carbon Dioxide; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CO2 (carbon dioxide) laser (Active Comparator): Patients randomized to this group will undergo CO2 laser excision of the sinus tracts in affected axilla
  Interventions: Procedure: CO2 (carbon dioxide) laser
- Surgical Deroofing (Active Comparator): Patients randomized to this group will undergo surgical deroofing of the sinus tracts in affected axilla
  Interventions: Procedure: Surgical Deroofing

INTERVENTIONS:
Procedure: CO2 (carbon dioxide) laser
  Arms: CO2 (carbon dioxide) laser
Procedure: Surgical Deroofing
  Arms: Surgical Deroofing

SUMMARY:
This study compares two well-known treatment options for Stage 2 hidradenitis suppurativa: carbon dioxide (CO2) laser excision versus surgical deroofing.

DETAILED DESCRIPTION:
* We will be treating patients with Stage 2 (interconnected sinus tracts and nodules) hidradenitis suppurativa who have somewhat active involvement (including drainage) in the axillae. We will only be treating ONE axilla per patient.
* After patients are screened and deemed appropriate candidates, they will be randomized to a treatment group: CO2 laser excision or surgical deroofing.
* For each patient, there will be a single intervention (either CO2 laser excision or surgical deroofing), after which there will be 5 planned follow-up appointment at following intervals: 1 week, 2 weeks, 4 weeks, 3 months, 6 months. This will take place over course of 6 months for each patient.
* During the study, subjects will be asked to provide information on quality of life measures, and filling out questionnaires (DLQI and Skindex29) at each visit.
* Inclusion criteria:

  1. Be at least 13 years old and have a diagnosis of hidradenitis affecting the underarms.
  2. Agree to follow and undergo all study-related procedures, and follow-up over six month period.
* Exclusion criteria:

  1. Patients who have already undergone surgical excision to affected area.
  2. Patients who are pregnant or breast feeding will not be able to take part in the study due to the unknown effects of CO2 laser in pregnant females, as well as risk of lidocaine use during pregnancy and breastfeeding
  3. Patients with a history of allergy to lidocaine or topical anesthetics will not be able to take part in this study.
  4. Patients with a history of vitiligo as the CO2 laser may cause new spots of depigmentation.
  5. Patients with a pacemaker/defibrillator in place.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 13 years old
2. Be otherwise healthy
3. Have a diagnosis of HS
4. Patients must have Hurley Stage II HS affecting the axilla, with one or more widely separated recurrent abscesses, with formation of a sinus tract and/or scarring
5. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form
6. Agree to follow and undergo all study-related procedures
7. If applicable, minors must have permission of legal guardian for participation in the study

Exclusion criteria:

1. Patients with HS Hurley stage I and III will be excluded from participation
2. Patients who are pregnant or breast feeding will not be able to take part in the study due to the unknown effects of CO2 laser in pregnant females, as well as risk of lidocaine use during pregnancy and breastfeeding
3. Any reason the investigator feels the patient should not participate in the study
4. If a patient misses ≥ 2 consecutive study visits, the patient will be excluded from further participation in this trial
5. History of allergy to lidocaine or topical anesthetics
6. Patients with a history of vitiligo as the CO2 laser may cause new spots of depigmentation
7. Patients with a pacemaker/defibrillator in place
8. Patients who have previously undergone surgical intervention and recurred in the axilla to be treated

Ages: 13 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2015-12-20 (Actual); Study Completion 2016-06-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life Measures | June 2014-February 2014
  Quality of Life measures will be measured via DLQI and Skindex29 patient surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States